CLINICAL TRIAL: NCT07145216
Title: Effect of Knack Pelvic Floor Contraction on Sexual Dysfunction in Females With Stress Urinary Incontinence
Brief Title: Effect of Knack Pelvic Floor Contraction on Sexual Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wafaa Ibrahim Hussein, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005672
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stress Urinary Incontinence (SUI); Sexual Dysfunction
MeSH Terms: conditions — Urinary Incontinence, Stress; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferential stimulation (Active Comparator): It will include 20 participants suffering from SUI associated with sexual dysfunction who will receive interferential stimulation for 20 minutes, 3 days per week for 8 weeks.
  Interventions: Other: Interfrential stimulation
- Interferential stimulation + Knack pelvic floor exercise (Experimental): It will include 20 participants suffering from SUI with sexual dysfunction who will receive interferential stimulation for 20 minutes in addition to the knack maneuver for 15 minutes, 3 days per week for 8 weeks.
  Interventions: Other: Interfrential stimulation; Other: Knack pelvic floor training

INTERVENTIONS:
Other: Interfrential stimulation — The participant will be positioned in semi-Fowler's position. Interferential therapy was given using the quadripolar method. Two electrodes were placed on the lower abdomen just above the outer half of the inguinal ligament, and another two on the inner aspect of the thigh near the origin of the adductor muscle. At the first treatment session, every participant will be examined for pelvic floor contraction by the finger palpation method using sterilized gloves to ensure the correct position of the electrodes. It will be set with intensity up to the tolerable limit of subjects, carrier frequency of 2000Hz, vector 900, rhythmic sweep frequency of 10-100Hz, and duration 20 minutes. Interferential therapy will be applied for the treatment procedure of all women in both groups for 20 minutes, 3days per week for 8 weeks.
Other: Knack pelvic floor training — The knack technique (Fitz et al., 2021):
  * The patient will be instructed to lie in supine lying position with flexed knees.
  * Ask the patient to contract the pelvic floor muscles for 2-4 seconds and relax for 4 seconds for 15 repetitions with 3 sets before and during coughing or sneezing .
  * Contract the PFM before and during all daily activities involving effort, before and during coughing, sneezing, laughing, walking up and down stairs, jumping, running, bending, lifting a weight from the floor, holding a child, pushing furniture to prevent urine leakage.
  * Contract PFM and hold for 2-4 seconds, relax 4 seconds, with 3 sets of 15 repetitions.
  Arms: Interferential stimulation + Knack pelvic floor exercise

SUMMARY:
This study aims to investigate the effect of knack pelvic floor contraction on sexual dysfunction in females with stress urinary incontinence.

DETAILED DESCRIPTION:
Stress urinary incontinence may have a tremendous effect on psychological and social well-being. Women with SUI report an inferior health-related quality of life (HRQOL) compared to continent women. Sexual well-being is an important aspect of women's health, and dysfunction can lead to a decrease in HRQOL and affect the marital relationship. It has been reported that women with UI also have problems with sexual activity. The presence of urinary leakage during intercourse can adversely affect sexual function.

Physiotherapy treatments for female SUI include PFMT such as knack maneuver, biofeedback, electrical stimulation, core stabilization, diet modifications, and behavioral therapy.

The knack is a simple, quick exercise technique that improves bladder control and increases PFM strength; it increases the urethral closure pressure, improves bladder stabilization and increases the structural support during PFM contraction. A previous study compared the knack effect on SUI using different methods like EMG biofeedback, verbal instructions, and vaginal palpation. It was found to have a positive impact on urinary symptoms, regardless of the teaching methods. Another previous study investigated the knack effect on vaginal laxity and found that it improved PFM contraction and sexual function and reduced vaginal laxity.

Up to now, no study has investigated the effect of the knack maneuver on female SUI associated with sexual problems, so this study will be the first one on this issue; therefore this study will be of valuable benefits and increase the knowledge of the physical therapist and health care provider in the women's health field.

ELIGIBILITY:
Inclusion Criteria:

1. Females with mild and moderate degrees of SUI according to Incontinence Severity Index score (mild: 1-2; and moderate: 3-4 scoring).
2. Their ages will range from 25 to 45 years old.
3. Their body mass index (BMI) will be less than 30 kg/m2.
4. They are multiparous women.
5. Females complain of sexual disorders related to SUI, identified by an FSFI score of less than 28.1
6. They have a sedentary lifestyle.

Exclusion Criteria:

1. Severe degree of SUI.
2. Other types of urinary incontinence, such as urge urinary incontinence and mixed urinary incontinence.
3. Other neurological diseases such as myasthenia gravis and Parkinsonism.
4. History of pelvic fractures.
5. Menopausal women.
6. Females with pelvic organ prolapse (POP).

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of pelvic floor muscle strength | 8 weeks
  PortablE biofeedback device will be used to assess pelvic floor muscle contraction. Each woman in both groups will be asked to count from 0 to 10 for 5 sets to achieve mental relaxation. Then, the area of the perineum will be cleaned with a disinfectant solution. The participant will insert the probe, which was covered with a condom and lubricated with hypoallergenic gel, into her vaginal cavity. The internal probe promotes proprioception and aids muscle awareness. The participants will be instructed to place the probe inside the vagina to a location where 0.5-1.0 cm of the probe is visible from the outside of the introitus. PFM strength will then be evaluated by a maximum voluntary contraction, as will be measured by squeeze pressure. Vaginal pressure testing will be performed with three repetitions of maximum voluntary contractions that each will be lasted for 3 s, with a 3-s rest between contractions. 2-minute rest break will then be taken, and the average score will be recorded.
Assessment of sexual function | 8 weeks
  The Arabic version of female sexual function Index score (FSFI) will be used to assess sexual function for all participating women in both groups before and after treatment program.
  All women in both groups will be asked to fill 5 domains of the questionnaire after explanation of them. The scoring system has a range of 2 to 36. According to Anis et al. (2011), a score above 28.1 indicated a good sexual life, whereas a score below 28.1 indicated reduced sexual function. The five categories of the questionnaire are severe (2-7.2), moderate (7.3-14.4), mild to moderate (14.5-21.6), mild (21.7-28.1 "cutoff point"), and no FSD (28.2-36)

SECONDARY OUTCOMES:
Assessment of symptoms of SUI | 8 weeks
  Incontinence Severity Index (ISI) will be used to assess SUI symptoms for all participating women in both groups before and after treatment program. All women in both groups will be asked to fill all items of questionnaire after a full explanation of them. The total score is the score for the first question multiplied by the score for the second question (0=dry, 1-2=slight, 3-4=moderate, 6-8=severe)
Assessment of quality of life | 8 weeks
  The world health organization quality of life questionnaire (WHOQOL) will be used to assess quality of life for all participating women in both groups before and after treatment. All women in both groups will be asked to fill all items of questionnaire after a full explanation of them.The score ranges from 0-20 indicating poor quality of life, 21-40 indicating moderate QOL, 41-60 indicating good QOL, and 61-80 indicating a very good QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A. Osman, PHD, Study Chair — Department of Women's Health, Faculty of Physical Therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt